CLINICAL TRIAL: NCT04149613
Title: Predictive and Prognostic Value of Inflammatory Markers and microRNA in Stage IV Colorectal Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Sally Temraz, Assistant Professor, American University of Beirut Medical Center
Other Study IDs: Bio-2018-0041
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer Stage IV
Keywords: biomarker; colorectal cancer; prognosis; prediction; microRNA; inflammation; dietary pattern
MeSH Terms: conditions — Colorectal Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample (Plasma) before treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal Cancer Patients: Newly diagnosed stage IV colorectal cancer patients
- Controls: cancer free

SUMMARY:
This study investigates the predictive and prognostic values of inflammatory markers and microRNA in stage IV colorectal cancer. The expression of inflammatory markers and microRNA in plasma will be correlated with tumor location, with dietary patterns and with survival during treatment.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is responsible for 10% of the world-wide cancer incidence and mortality. Recent data have shown that tumors arising from different regions of the colon differ in their molecular characteristics which causes translate into a differential clinical outcome.Several studies described the role of microRNA expression in the initiation and progression of CRC and its response to different therapeutic strategies. Other studies have shown that systemic inflammation is a key determinant role of clinico-pathological outcomes in patients with CRC. We therefore aim to evaluate the expression of selected microRNA and inflammatory markers in patients with stage IV colorectal cancer and assess their correlation with tumor location, dietary patterns, survival rates, response to systemic chemotherapy and other clinic-pathological parameters. We believe that identifying a predictive and prognostic panel made up of circulating microRNA and inflammatory markers may perhaps explain the difference in outcome between right and left colon and perhaps impact the clinical practice in patients with stage IV colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Stage IV colorectal cancer
2. Treatment naïve
3. For the control group: adult individuals (above 18 years) with no cancer disease

Exclusion Criteria:

Any disease or condition that may alter the inflammatory and immune status of subjects at baseline, such as:

1. Diagnosis of inflammatory bowel disease such as ulcerative colitis and crohn's disease.
2. Diagnosis of active systemic autoimmune disease
3. Chronic / recent use of corticosteroids
4. Use of immunosuppressant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary physicians will identify patients who are treatment naïve, stage IV colorectal cancer patients, and exclude the patients, who have a history of an inflammatory bowel disease, or an active systemic autoimmune disease, and who have a chronic / recent use of corticosteroids or on immunosuppressant drugs therapy. Recruitment will be done for patients admitted to the chemotherapy infusion unit at the Naef K. Basile Cancer Institution at the American University of Beirut Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Level of inflammatory markers | At diagnosis before chemotherapy
  Level of C-reactive protein (CRP), Erythrocyte sedimentation rate (ESR), serum albumin, fibrinogen, haptoglobin, lymphocyte monocyte ratio (LMR), neutrophil lymphocyte ratio (NLR) and platelets lymphocytes ratio (PLR)
microRNA expression Level | At diagnosis before chemotherapy
  miR-21, miR-19a, miR-155, miR-200c, miR-210, miR-126, miR-345, miR-31, miR-29a, miR-200b, and miR-203

SECONDARY OUTCOMES:
Dietary pattern | At diagnosis before chemotherapy and every 3 months
  Associations of dietary patterns (such as the Mediterranean diet and DII) with inflammatory markers, and microRNA expression

CONTACTS AND LOCATIONS:
Overall Officials: Sally Temraz, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon